CLINICAL TRIAL: NCT03118700
Title: Postexercise Central Blood Pressure and Hemodynamic Response After Continuous and Aerobic Interval Exercise
Brief Title: Central Hemodynamic Exercise Responses Study
Acronym: CHeER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Researcher left
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: CHeER
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Exercise; Central Blood Pressure
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-exercise Control (No Intervention): Subjects will come to the laboratory for 4 hours and their blood pressure will be measured every 10 minutes using the Oscar 2 with SphygmoCor ambulatory blood pressure system, and cardiac output will be measured with 10-second averages using the PhysioFlow. During this time, subjects will remain seated with their body posture maintained constant
- Aerobic Interval Exercise (Experimental): Subjects will be equipped with a heart rate (HR) monitor and perform an interval exercise bout on a cycle ergometer. To warm up, subjects will cycle at a work rate associated with 50% HRmax for 10 minutes. Wattage will then increase and subjects will do four 4-minute intervals at a work rate associated with 90%-95% HRmax, separated by 3 minutes of active recovery at a work rate associated with 50% HRmax. Subjects will be given a 5-minute cool-down period at a work rate associated with 50% HRmax. After the exercise, subjects will remain seated in the lab for 4 hours and their blood pressure will be measured every 10 minutes using the Oscar 2 with SphygmoCor ambulatory blood pressure system, and cardiac output will be measured with 10-second averages using the PhysioFlow.
  Interventions: Other: Aerobic Interval Exercise
- Continuous Exercise (Experimental): Subjects will be equipped with a heart rate (HR) monitor and perform an interval exercise bout on a cycle ergometer. To warm up, subjects will cycle at a work rate associated with 50% HRmax for 10 minutes. Wattage will then increase and subjects will perform a 30-minute exercise bout at a HR that elicits 75%-80% of their measured HRmax. Work rate will be adjusted, if needed, to keep HR within this value. Subjects will be given a 5-minute cool-down period at a work rate associated with 50% HRmax. After the exercise, subjects will remain seated in the lab for 4 hours and their blood pressure will be measured every 10 minutes using the Oscar 2 with SphygmoCor ambulatory blood pressure system, and cardiac output will be measured with 10-second averages using the PhysioFlow.
  Interventions: Other: Continuous exercise

INTERVENTIONS:
Other: Aerobic Interval Exercise — Subjects will perform an interval exercise bout on a cycle ergometer. To warm up, they will cycle at a work rate associated with 50% of their max heart rate (HR) for 10 minutes. Wattage will then increase and they will do four 4-minute intervals at a work rate associated with 90%-95% HRmax, separated by 3 minutes of active recovery at a work rate associated with 50% HRmax They will be given a 5-minute cool-down period at a work rate associated with 50% of their max HR. After the exercise, they will remain in the lab for 4 hours and their blood pressure will be measured every 10 minutes using an automated blood pressure monitor and cardiac output will be measured using the PhysioFlow. They will remain seated during this time
  Arms: Aerobic Interval Exercise
Other: Continuous exercise — Subjects will perform a 30-minute continuous exercise bout on a cycle ergometer. To warm up, they will cycle at a work rate associated with 50% of their max heart rate (HR) for 10 minutes. Wattage will then increase and they will perform a 30-minute exercise bout at a work rate associated with 75%-80% of their max HR. They will be given a 5-minute cool-down period at a work rate associated with 50% of their max HR. After the exercise, they will remain in the lab for 4 hours and their blood pressure will be measured every 10 minutes using an automated blood pressure monitor and cardiac output will be measured using the PhysioFlow. They will remain seated during this time.
  Arms: Continuous Exercise

SUMMARY:
The purpose of this study is to examine the acute effect of continuous and aerobic interval exercise on postexercise central BP response in men with an elevated blood pressure.

DETAILED DESCRIPTION:
The specific aim of this study is to compare postexercise central blood pressure after continuous and aerobic interval exercise. It is hypothesized that aerobic interval exercise will produce a longer duration postexercise hypotensive response compared to continuous exercise. 14 healthy, inactive (defined as less than 60 minutes of moderate to vigorous physical activity per week, as characterized by accelerometry) men aged 18-45 yr, who have high normal BP or stage 1 hypertension (systolic BP (SBP) 120-159 mmHg or diastolic BP (DBP) 80-99 mmHg) according to JNC 8 established guidelines, will be included in this randomized cross-over design study. Each subject will complete three conditions in a randomized order: aerobic interval exercise, continuous exercise, and non-exercise control.

For the aerobic interval exercise condition, subjects will be equipped with a heart rate (HR) monitor and asked to perform an interval exercise bout on a cycle ergometer. To warm up, subjects will cycle at a work rate associated with 50% HRmax for 10 minutes. Wattage will then increase and subjects will do four 4-minute intervals at a work rate associated with 90%-95% HRmax, separated by 3 minutes of active recovery at a work rate associated with 50% HRmax. Subjects will be given a 5-minute cool-down period at a work rate associated with 50% HRmax. After the exercise, subjects will remain in the lab for 4 hours and their blood pressure will be measured every 10 minutes using the Oscar 2 with SphygmoCor ambulatory blood pressure system, and cardiac output measured in 10-second averages using the PhysioFlow. During this time, subjects will remain seated with their body posture maintained constant.

For the continuous exercise condition, subjects will be equipped with a HR monitor and asked to perform a continuous exercise bout on a cycle ergometer. To warm up, subjects will cycle at a work rate associated with 50% HRmax for 10 minutes. Wattage will then increase and subjects will perform a 30-minute exercise bout at a HR that elicits 75%-80% of their measured HRmax. Work rate will be adjusted, if needed, to keep HR within this value. Subjects will be given a 5-minute cool-down period at a work rate associated with 50% HRmax. After the exercise, subjects will remain in the lab for 4 hours and their blood pressure will be measured every 10 minutes using the Oscar 2 with SphygmoCor ambulatory blood pressure system, and cardiac output measured in 10-second averages using the PhysioFlow. During this time, subjects will remain seated with their body posture maintained constant.

For the non-exercise control condition, subjects will be asked to come to the laboratory for 4 hours and have their blood pressure will be measured every 10 minutes using the Oscar 2 with SphygmoCor ambulatory blood pressure system, and cardiac output measured in 10-second averages using the PhysioFlow. During this time, subjects will remain seated with their body posture maintained constant.

ELIGIBILITY:
Inclusion Criteria:

* Inactive (defined as less than 60 minutes of moderate to vigorous physical activity per week, as characterized by accelerometry) non-smoking men who have high normal blood pressure or stage 1 hypertension (systolic BP (SBP) 120-159 mmHg or diastolic BP (DBP) 80-99 mmHg) according to JNC 8 established guidelines

Exclusion Criteria:

* Men over 45 years old, who register more than 60 minutes/week of moderate-to-vigorous physical activity, or have a blood pressure less than 120/80 mmHg will be excluded. Those who answer positively (i.e., yes) on The Physical Activity Readiness Questionnaire (PAR-Q) will be excluded from participating in the study. Those with known cardiovascular, pulmonary, renal or metabolic disease, or having symptoms suggestive of these diseases will be excluded from the study as per current American College of Sports Medicine guidelines. Current smokers or anyone with contraindications to vigorous exercise will be excluded from the study as well. Subjects on medications used for the treatment of symptomatic cardiovascular disease will be excluded

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Postexercise central blood pressure response after aerobic interval and continuous exercise | 4 hours
  After the subject performs both an aerobic interval and continuous exercise, blood pressure will be measured every 10-minutes using an ambulatory blood pressure monitor

SECONDARY OUTCOMES:
Postexercise hemodynamic response after aerobic interval and continuous exercise | 4 hours
  After the subject performs both an aerobic interval and continuous exercise, cardiac output will be measured in 10-second averages using the PhysioFlow

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No